CLINICAL TRIAL: NCT04837690
Title: The Use of Underwater Endoscopic Mucosal Resection for Medium-sized Pedunculated Colon Polyps: A Prospective Observational Study
Brief Title: UEMR for Medium-sized Pedunculated Colon Polyps
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AUEMR-1.0
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Colon Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UEMR
  Interventions: Procedure: UEMR

INTERVENTIONS:
Procedure: UEMR — (1) the colorectal lumen was completed deflated with 500-1000 mL sterile water using a flushing pump; (2) the lesion and 2-3 mm of normal mucosa surrounding the base of the polyp were snared and subsequently resected with an electrosurgical generator

SUMMARY:
Underwater EMR (UEMR) is an emerging technique for endoscopic resection. The purpose of this research is to observ wether the UEMR for medium-sized pedunculated polyps is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

Patients age between 18-75 years old with pedunculated colonic polyps (measuring between 10 and 20mm), who willing to participate in this study.

Exclusion Criteria:

1. pregnancy,
2. inflammatory bowel disease,
3. familial polyposis
4. the use of anticoagulant therapy or antiplatelet therapy
5. the absence of informed patient consent.
6. Polyps showing signs of deep submucosal invasion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients or inpatients requiring polypectomy
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
The rate of bleeding | 1 Day of colonoscopy
  the bleeding was defined as the active hemorrhage lasted for ≥ 30 s or other condition requires immediate intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China